CLINICAL TRIAL: NCT03672877
Title: Randomized Controlled Trial of Early Intensive Leg Exercise to Improve Walking in Children With Diplegia From Encephalopathy of Prematurity
Brief Title: Randomized Controlled Trial of Early Intensive Leg Exercise to Improve Walking in Children With Diplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00080569
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Spastic Diplegia; Periventricular Leukomalacia
Keywords: Physical Therapy; Rehabilitation; Walking
MeSH Terms: conditions — Cerebral Palsy; Leukomalacia, Periventricular

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive 3 months of intervention immediately (Immediate Group) or to be observed for 6 months (Delay Group). Participants in the Delay Group will be offered the intervention once the observation period is complete.
Who Masked: Outcomes Assessor
Masking Description: Physical therapy assessors will be blinded to the child's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate training group (Experimental): Children will participate in intensive exercise intervention for 3 months and will be followed for 9 months following the intervention
  Interventions: Behavioral: Intensive exercise
- Delay training group (No Intervention): Children will be assessed for 6 months with no intervention. After the 6 month period children will be given the same intervention as the immediate group and followed for 3 months after the intervention.

INTERVENTIONS:
Behavioral: Intensive exercise — Intensive, child-initiated activities of the lower extremities including walking (with or without support), kicking, jumping, standing balance, climbing stairs and slopes and other leg activities. Small weights will be added to the ankle and foot to increase the intensity of the exercise. Sessions will be one hour long, 4 days a week. A physical therapist or designate will supervise sessions.
  Arms: Immediate training group

SUMMARY:
This is a randomized controlled trial, comparing 3 months of intensive leg exercise to standard physiotherapy care for the improvement of gross motor function in young children with spastic diplegia.

DETAILED DESCRIPTION:
Children born prematurely are at risk of brain injury that can result in cerebral palsy, most often affecting both legs. Current treatment is largely passive, including leg braces, repeated injection of a paralyzing agent (botulinum toxin) in muscles that are abnormally active, and surgery as deformities occur. Active, physical therapy for weak muscles is infrequent, occurring twice a month or less. Yet, recent work in mammals show that early brain injury can be alleviated by intensive exercise therapy, but only while the animal is very young.

Building on our success with early, intensive therapy for children with perinatal stroke, we will apply intensive therapy for the legs in children with cerebral palsy involving both legs. Children (8 mo - 3 yr old) will be randomly assigned to start treatment immediately or delay treatment for 6 months. The delay period controls for improvement without treatment. The children in the Delay Group will have the option to receive the same treatment after the delay period. The therapy will be guided by physical therapists, and centered on play. Measures will be taken before, during and after the delay and treatment periods. Measures will include clinical scores of motor development, proficiency of walking, participation at home, and physiological measures of motor and sensory function. All children will be followed until they turn 4 yr old, to determine if there are long term benefits. The cost-effectiveness of the intervention will be evaluated by a health economist. We anticipate that early intensive exercise will improve mobility, facilitate earlier and better walking, and that the effects will be enduring.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral motor impairment of the lower extremities
* Periventricular white matter injury from encephalopathy of prematurity
* Able to stand with some support

Exclusion Criteria:

* Substantial upper extremity involvement - Manual Abilities Classification System (MACS) Level ≥3
* Uncontrolled epilepsy or infantile spasms in the past 6 months
* Cardiovascular or musculoskeletal complications that preclude participation in intensive exercise
* Botulinum toxin-A (BTX-A) injections in the legs in the last 6 months

Ages: 8 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Functional Measure - 66 Items (GMFM-66) | From Baseline to 6 months
  This is a 66 item criterion-referenced observational measure to assess change in gross motor function of children with cerebral palsy.

SECONDARY OUTCOMES:
Change on Pediatric Quality of Life Measure module for cerebral palsy (PedsQL CP) | From Baseline to 6 months
  A questionnaire format completed by parents including 5 scales: 1) daily activities, 2) movement and balance, 3) pain and hurt, 4) fatigue, and 5) eating activities.
Change in stiffness at the ankle | From Baseline to 6 months
  The portable spasticity assessment device (PSAD) will be used to measure response to stretch in the ankle plantarflexors. A hand-held segment of the device is applied to a limb segment to measure the forces applied by the hand to the limb and the motion of the limb. Disposable, surface electromyographic electrodes are applied to the skin of the limb to measure the muscle activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie Yang, Phd, Principal Investigator — Universtiy of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta